CLINICAL TRIAL: NCT01243190
Title: Ofatumumab Early Treatment for High-Risk Treatment-Naive, Early Stage (0-II) Patients With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: Ofatumumab for High-Risk Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0241; NCI-2011-00745 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-11-12; First posted 2010-11-18 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: leukemia; small lymphocytic leukemia; SLL; CLL; ofatumumab; untreated; early stage; high-risk
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Loading dose 300 mg by vein on Day 1 of Cycle 1; and full dose 1000 mg over 4 hours 1 time each week for 7 additional weekly doses (8 doses).
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Loading first dose 300 mg by vein on Day 1 of Cycle 1; and full dose 1000 mg over 4 hours 1 time each week for 7 additional weekly doses (8 doses).
  Other Names: Arzerra

SUMMARY:
The goal of this clinical research study is to learn if ofatumumab can help to control CLL/SLL that has not yet been treated. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Ofatumumab is designed to bind to the surface of some of the white blood cells (B-cells). It may destroy cancer cells that come from B-cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive a "loading dose" (a lower dose given first, to lower the risk of a bad reaction to the study drug) of ofatumumab by vein on Day 1 of Cycle 1. The loading dose is less than one-third (1/3) of the normal dose. You will then receive the normal dose over 4 hours 1 time each week (+/- 3 days). The doses may be given more slowly, if your doctor thinks it is needed. All doses of the study drug will be given at M. D. Anderson.

Benadryl (diphenhydramine) and glucocorticoids (steroids such as prednisolone) will be given by vein 30 minutes to 2 hours before you receive ofatumumab to help prevent side effects. You will also take pills of acetaminophen (Tylenol) to help prevent side effects. If no side effects occur, these "pre-medications" may be reduced or not given after the second infusion.

Study Visits:

One (1) time each week, before you receive ofatumumab:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about how you are feeling, about any side effects you may be having, and about any changes in your health since the last visit.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Length of Study:

You may continue taking the study drug until Day 50, as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, if you develop hepatitis B, or if you decide to go off study.

End-of-Treatment Visit:

On the day of your last treatment or after you stop receiving the study drug for any reason, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about how you are feeling, about any side effects you may be having, and about any changes in your health since the last visit.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for hepatitis testing.

Follow-Up:

About 3 months (+/- 2 weeks) after the end-of-treatment visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about how you are feeling, about any side effects you may be having, and about any changes in your health since the last visit.
* You will have a bone marrow aspirate and biopsy, as well as CT scans of the chest, abdomen, and pelvis, to check the status of the disease.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for hepatitis testing.

Every 3 months (+/- 4 weeks) after the end-of-treatment visit for 6 months:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about how you are feeling, about any side effects you may be having, and about any changes in your health since the last visit.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for hepatitis testing.

Every year (+/- 4 weeks) after the end-of-treatment visit:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about how you are feeling, about any side effects you may be having, and about any changes in your health since the last visit.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspirate and biopsy, as well as CT scans of the chest, abdomen, and pelvis, to check the status of the disease.

This is an investigational study. Ofatumumab is FDA approved and commercially available for use in the treatment of CLL. The use of ofatumumab as an early treatment for patients with CLL/SLL who have not received other treatment is investigational.

Up to 44 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic lymphocytic leukemia (CLL)/ small lymphocytic leukemia (SLL), previously untreated, Rai stage 0-ll
2. At least 1 of the following high-risk features for previously untreated patients: Rai stage II disease; Rai stage 0-I with disease-related fatigue; Serum beta2M >/= 3 mg/L; Absolute lymphocyte count >/= 25,000/uL; Unmutated IGHV gene or IGHV3-21; ZAP70 positive (>/= 20% by flow cytometry or positive by immunohistochemistry); CD38 positive (>/= 30% by flow cytometry); OR Deletion 11q or 17p by FISH
3. ECOG PS </= 2
4. Age >/= 18 years
5. Patients must have adequate renal and hepatic function (creatinine <2mg/dL, total bilirubin <2mg/dL). Patients with renal or liver dysfunction due to organ infiltration with CLL may be eligible after discussion with the study chairman
6. Provide informed consent
7. Female patients (including those < 1 year post-menopausal) and male patients who have not undergone previous surgical sterilization must agree to use contraception.

Exclusion Criteria:

1. Presence of 2008 IWCLL/NCI-WG indication for CLL treatment: Constitutional symptoms related to CLL/SLL: Fever > 100.5 degrees F for >/= 2 weeks or night sweats for > 1 mo, both without evidence of infection; Unintentional weight loss of >/= 10% body weight in previous 6 months; Extreme fatigue (ECOG PS > 2; inability to work or perform usual activities); Lymphocyte doubling time of </= 6 months or 50% increase in absolute lymphocyte count within 2 months; Progressive anemia (Rai stage III) or thrombocytopenia (Rai stage IV); Recurrent infections unrelated to hypogammaglobulinemia; Autoimmune phenomenon poorly responsive to corticosteroids or other standard therapy; Massive, progressive or symptomatic lymphadenopathy (> 10 cm in longest diameter) or splenomegaly (> 6 cm below left costal margin)
2. Prior or concurrent chemotherapy, radiotherapy, or immunotherapy for CLL
3. Active infection (febrile and requiring IV/PO antibiotics), including hepatitis C or HIV, or significant medical illness including renal, cardiac, pulmonary disease, or current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
4. Positive serology for Hepatitis B virus (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the patient will be excluded. -- Consult with a physician experienced in care and management of subjects with hepatitis B to manage/treat subjects who are anti-HB positive.
5. Pregnant or breast feeding females are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Weirda, BS,MD,PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ofatumumab
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 59 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 38
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response (CR)
Description: 2008 International Workshop on CLL (IWCLL) update of the National Cancer Institute-sponsored Working Group (NCI-WG) outlined specific criteria of Complete Response (CR) for diagnosing CLL. CR is defined as Marrow normocellular, no CLL cells, no B-lymphoid nodules, hemoglobin of ≥11.0 g/dL (untransfused and without erythropoietin), Platelet count of ≥100 × 10^9/L, circulating lymphocyte count normal, no constitutional symptoms, Liver and/or spleen size <13 cm; liver size normal, lymph nodes ≥ 1.5 cm.
Time Frame: Up to 12 years
Population: Of the 44 participants registered, 43 were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 43
Participants | 11

ADVERSE EVENTS:
Time Frame: Up to 12 years
Arm/Group | Ofatumumab
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 22/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab (N=44)
INFUSION REACTION (Investigations) | 21 (21)
AUTOIMMUNE HEPATITIS (Immune system disorders) | 1 (1)
ELEVATED AST (Investigations) | 1 (1)
LIVER BX (Surgical and medical procedures) | 1 (1)
RADIATING LEG PAIN (General disorders) | 1 (1)
SHINGLES (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab (N=44)
Hypertension (Vascular disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 11 (11)
cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 4 (4)
fatigue (General disorders) | 32 (32)
headache (Nervous system disorders) | 5 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (7)
Back Pain (General disorders) | 3 (3)
Neck Pain (General disorders) | 4 (4)
Stoma pain (Gastrointestinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 27 (27)
Neutropenia (Blood and lymphatic system disorders) | 17 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (25)
Lymphocytes (Investigations) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT01243190/Prot_SAP_000.pdf